CLINICAL TRIAL: NCT00510653
Title: A Phase II Study of Gleevec in Patients With Recurrent Platinum-Resistant, Taxane-Resistant Epithelial Ovarian Cancer, Primary Peritoneal Cancer, or Fallopian Tube Cancer
Brief Title: Gleevec Study for Patients With Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID01-707
Record Dates: First submitted 2007-07-31; First posted 2007-08-02 (Estimated); Results first posted 2013-08-23 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-06

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Primary Peritoneal Cancer; Fallopian Tube Cancer; Recurrent Platinum-Resistant; Taxane-Resistant; Epithelial Ovarian Cancer; Imatinib Mesylate; Gleevec; STI571; Protein tyrosine kinase inhibitor
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imatinib Mesylate (Experimental): 600 mg/day orally for 6 Weeks
  Interventions: Drug: Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib Mesylate — 600 mg by mouth daily for 6 Weeks
  Other Names: Imatinib; Gleevec; STI571; NSC-716051

SUMMARY:
Primary Objectives:

1. To determine the efficacy of Gleevec in patients with recurrent platinum-resistant, taxane-resistant epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer whose tumor expresses either c-KIT, platelet-derived growth factor receptor (PDGRF), or ABL.
2. To determine the nature and degree of toxicity of Gleevec in this cohort of patients.

DETAILED DESCRIPTION:
Imatinib Mesylate is a new medication that blocks several proteins important in the development of cancer. Before going on study, potential participants will have their tumor tested for c-KIT, PDGFR, and ABL for positivity. Those participants who have at least one positive biomarker will be eligible for treatment.

Before treatment starts, participants will have a complete checkup, blood tests, chest x-ray, and heart function test. Women able to have children must have a negative blood pregnancy test. A blood sample (3 teaspoons) will be taken once a week during treatment and at the end of treatment. A complete exam will also be done at the end of treatment. Tumors will be measured by computed tomography (CT) scan every 6 weeks while one study and at the end of treatment.

Participants in this study will take Imatinib Mesylate by mouth in a single dose on a daily basis. Participants will be treated for 6 weeks, which is one cycle of therapy. After 6 weeks, participants will be evaluated for side effects and tumor response. The dose may be decreased for the next cycle if participants side effects. Participants will be removed from the study if the tumor gets worse. Participants may remain on the study as long as the tumor has not gotten worse and there are no intolerable side effects.

This is an investigational study. Imatinib Mesylate has been approved for chronic myelogenous leukemia patients. However this is an investigational study of Imatinib Mesylate in patients with ovarian, tubal, or peritoneal cancer. Participants may responsible for the cost of all or part of this drug. At least 24 and as many as 74 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic epithelial ovarian, primary peritoneal cancer, or fallopian tube cancer previously treated with a platinum/taxane-containing regimen. Patients may have either low-grade or high-grade recurrent epithelial tumors.
2. Patients with high-grade tumors must be platinum/taxane resistant, as defined by: progression of disease while on a first-line platinum/taxane regimen or tumor progression within 6 months of completion of a platinum/taxane regimen.
3. Patients with high-grade tumors may have failed no more than 4 prior chemotherapy regimens. All taxane/platinum therapies will be counted as one regimen.
4. Patients with low-grade tumors may have failed unlimited prior therapies.
5. Patients' tumor tissue must express one or more of the following biomarkers: c-KIT, PDGFR or ABL. Positivity will be defined as 2+ or 3+ on immunohistochemical staining.
6. All patients must have measurable disease. Measurable disease is defined as lesions which can be measured by physical examination or by means of imaging techniques. Ascites and pleural effusions are not to be considered measurable disease. An elevated serum CA 125 level without associated measurable tumor is not to be considered measurable disease.
7. Patients must have a pretreatment granulocyte count (i.e., segmented neutrophils + bands) of > 1,500/Fl, a hemoglobin level of = 9.0 gm/dL and a platelet count of > 100,000/Fl.
8. Patients must have adequate renal function as documented by a serum creatinine <2.0 mg/dL.
9. Patients must have adequate hepatic function as documented by a serum bilirubin <1.5 mg/dL, regardless of whether patients have liver involvement secondary to tumor. Aspartate transaminase (SGOT) must be < 3* institutional upper limit of normal unless the liver is involved with tumor, in which case the aspartate transaminase must be < 5* institutional upper limit of normal.
10. Patients must have an estimated life expectancy of 12 weeks or greater.
11. Zubrod performance status of 0, 1, or 2.
12. Patients must be older than age 18.
13. Patients must have signed an approved informed consent.

Exclusion Criteria:

1. Patients who have previously received Gleevec.
2. Patients with any active or uncontrolled infection, including known HIV infection.
3. Patients with psychiatric disorders that would interfere with consent or follow-up.
4. Patients with a history of myocardial infarction within the previous six months or congestive heart failure requiring therapy.
5. Patients with a history of prior malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for at least five years.
6. Pregnant or lactating women. Men and women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
7. Presence of clinically apparent central nervous system metastases or carcinomatous meningitis.
8. Patients with a history of seizures are ineligible. Patients receiving phenytoin, phenobarbital, or other antiepileptic prophylaxis are ineligible.
9. Patients with any other severe concurrent disease which in the judgment of the investigator, would make the patient inappropriate for entry into this study, including significant hepatic, renal, or gastrointestinal diseases.
10. Patients with a deep venous or arterial thrombosis (including pulmonary embolism) within 6 weeks of study entry.
11. Patients who are receiving warfarin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2002-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Gershenson, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 7, 2002 to September 30, 2009. All registration was done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of the 73 enrolled, 27 were excluded as not eligible and one inevaluable for the study. Another four (4) participants were found to be not eligible following screening.
Period: Overall Study
Arm/Group | Imatinib Mesylate
Started | 24
Completed | 13
Not Completed | 11
Not completed — Withdrawal by Subject | 8
Not completed — Monetary | 3

BASELINE CHARACTERISTICS:
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 24
Age Continuous [Median (Full Range); unit: years] | 52 [32 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR = participant proportion with responsive disease: Complete Response (CR): disappearance all clinically detectable malignant disease for at least 4 weeks, no new lesions; Partial Response (PR): >/= 50% decrease sum of products of perpendicular diameters of all measurable lesions for at least 4 weeks; Stable Disease: does not qualify for CR, PR or progression. Progressive Disease: a 25% or > increase in sum of products of measurable lesions over smallest sum observed, OR reappearance of lesion which had disappeared, OR appearance of new lesion/site. Response determined every 6 week cycle.
Time Frame: 6 weeks with re-evaluation every 6 weeks or until disease progression
Population: Two participants were not evaluable for response: in 1 participant, early toxicity caused discontinuation of the drug, and the other patient had an intestinal obstruction requiring palliative surgery after 1 day of therapy.
Measure: Number; unit: participants
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 11
participants
  Complete Response | 0
  Partial Response | 0

ADVERSE EVENTS:
Time Frame: 7 years
Arm/Group | Imatinib Mesylate
Serious Adverse Events (participants affected / at risk) | 4/13
Other Adverse Events (participants affected / at risk) | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib Mesylate (N=13)
Granulocytopenia (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 1
Febrile neutropenia (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib Mesylate (N=13)
Fatigue (General disorders) | 8
Nausea-vomiting (Gastrointestinal disorders) | 8
Edema (Vascular disorders) | 5
Neuropathy (sensory) (Nervous system disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 5
Weight Gain (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No